CLINICAL TRIAL: NCT00800449
Title: Prospective Assessment of the Distribution of Haptoglobin Phenotype in Septic and Non Septic Pre-term Neonates (PTSH)
Brief Title: Distribution of Haptoglobin Phenotype in Septic and Non Septic Pre-term Neonates (PTSH)
Status: Completed | Type: Observational
Sponsor: Irina Kessel (Other)
Collaborators: Carmel Medical Center (Other); Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Irina Kessel, MD, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Other Study IDs: PTSH001
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Neonatal Sepsis
Keywords: Haptoglobin; sepsis; premature babies
MeSH Terms: conditions — Neonatal Sepsis; Sepsis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hp phenotype in blood test.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Haptoglobin (Hp) gene locus at chromosome 16q22 is polymorphic with two alleles denoted 1 and 2 .The gene product exists in three phenotypes: 1-1, 2-1, and 2-2.

The Haptoglobin 2 allele is found only in man and is believed to have arisen from the Haptoglobin 1 allele by a partial intragenic duplication. Haptoglobin 2 allele frequency is higher than the Haptoglobin 1 allele. It has been hypothesized that the Haptoglobin 2 allele was spread in man due to its selective advantage against life-threatening infections.

In vitro, only the Haptoglobin 2 allele protein, binds to the streptococcus T antigen, resulting in its aggregation and slowing its growth .

Individuals homozygous for the Haptoglobin 1 allele (1-1 genotype) are more prone to the streptococcal infection than individuals with the Haptoglobin 2 allele(2-1 or 2-2 genotype).

The investigators wish to explore the linkage between Hp phenotype and sepsis in pre-term neonates, considering that in this early stage in life, genetic properties which provide a defense against infectious agents will be of heightened importance.

DETAILED DESCRIPTION:
The Haptoglobin (Hp) gene locus at chromosome 16q22 is polymorphic with two alleles denoted 1 and 2 .The gene product exists in three phenotypes: 1-1, 2-1, and 2-2. Hp 2 allele DM individuals have larger myocardial infarctions than homozygous Hp 1 DM individuals. This may be due to differences in the antioxidant and anti-inflammatory properties of these proteins.The same phenomenon was demonstrated in a murine coronary ischemia-reperfusion model.

The Haptoglobin is an acute phase protein with anti-oxidant, bacteriostatic and anti-inflammatory functions.

The Haptoglobin 2 allele is found only in man and is believed to have arisen from the Haptoglobin 1 allele by a partial intragenic duplication. Haptoglobin 2 allele frequency is higher than the Haptoglobin 1 allele. It has been hypothesized that the Haptoglobin 2 allele was spread in man due to its selective advantage against life-threatening infections.

In vitro, only the Haptoglobin 2 allele protein, binds to the streptococcus T antigen, resulting in its aggregation and slowing its growth .

We proposed that in individuals homozygous for the Haptoglobin 1 allele (1-1 genotype), the streptococcal infection would be more severe than in individuals with the Haptoglobin 2 allele (2-1 or 2-2 genotype).

During a severe outbreak of impetigo in two infantry units in the Israeli Defense Forces, over 60% (57/91) of the soldiers developed impetigo caused by a single pathogen-group A streptococcus. 33% of them developed serious life-threatening complications requiring hospitalization. The risk of Haptoglobin 1-1 genotype individuals developing severe infection was significantly higher than individuals with Haptoglobin 2 genotype (45.5% (5/11) vs. 17.5% (14/80), risk ratio 2.6 (95% confidence interval 1.2-5.8), p=0.05). This supports the notion that the Haptoglobin genotype determines the susceptibility to streptococcus infection, an important pathogen early in human evolution, and explains the spread of Haptoglobin 2 allele in human.

Another study demonstrated that Diabetic dialysis patients at the age of 60 and above carrying the Hp1-1 phenotype had a lower mortality rate compared to the patients who are Hp2-2. However, younger population has shown the opposite. This can be explained by the survivorship pattern of Hp1-1 diabetic patients who have lower risk for diabetic complications. They will also survive dialysis in older age by suffering less from vascular complications compared to Hp2-2. However, in Hp2-2 younger patients, the infectious parameter is more significant and mortality will be lower.

We wish to explore the linkage between Hp phenotype and sepsis in pre-term neonates, considering that in this early stage in life, genetic properties which provide a defense against infectious agents will be of heightened importance.

During the study period of one year, all preterm neonates (a total of 150 preterm babies, 35 weeks or younger) admitted to the preterm unit at Carmel hospital will be typed for Hp phenotype by a blood test. Hp phenotyping needs only about 500 microliters of blood which will be taken during routine blood drawn. All blood samples will be identified with the patient's I.D. number and name in addition to the study consecutive serial number. The blood samples will be sent to the laboratory of vascular medicine in the faculty of medicine at the Technion. If the number of participating infants during one year will be insufficient (less than 150), we will ask for additional permission of the ethical committee to continue the study for the second year.

Septic neonates will be recognized by clinical deterioration (abnormal body temperature and/or disturbed skin perfusion and/or apathy and/or increase in apnea/bradycardia episodes and/or abnormal CBC, leukocytosis or leucopenia or left shift or thrombocytopenia) and concomitant positive blood cultures, without another explanation of non infectious etiology. Details of the bacteria including antibiotic resistance profile will be documented. Demographic data will be collected for all patients.

In addition data regarding known pre-maturity complications such as Retinopathy of Pre-maturity (ROP), Necrotizing Entero-Colitis (NEC), Broncho-Pulmonary Dysplasia (BPD) will be assessed and documented according to the admission summary.

Blood transport, Hp typing and data collection will be done by a MD student as part of her MD thesis.

As part of the informed consent, we will ask the permission for a possible follow up one year after discharge from the hospital which will be done by a phone questionnaire and acquiring the patients medical file data with the help of his family

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies born at 35 week gestational age and younger being admitted to the preterm unit in Carmel Medical Center over a period of one year.

Exclusion Criteria:

* Pre-term neonates with serious congenital defects.

Ages: 24 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm neonates ( a total of 150 preterm babies, 35 weeks or younger) admitted to the NICU in Carmel hospital.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irena Kessel, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel